CLINICAL TRIAL: NCT07117903
Title: Zhongshan Ketogenic Diet Study 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhiyong Qi, Dr., Fudan University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Y2024-146
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Platelet Function and Thrombus Formation
MeSH Terms: interventions — Aspirin; Diet, Ketogenic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Normal diet + vehicle — Participants in the control group were instructed to maintain their usual diet for the duration of the study. While they were free to choose their food, they were required to provide a detailed dietary record. After diet intervention, whole blood will be drawn and incubated with vehicle drug.
Dietary Supplement: Normal diet + aspirin — Participants in the control group were instructed to maintain their usual diet for the duration of the study. While they were free to choose their food, they were required to provide a detailed dietary record. After diet intervention, whole blood will be drawn and incubated with aspirin.
Dietary Supplement: Ketogenic diet + vehicle — The calorie-restricted KD intervention consisted of a very-low-carbohydrate, high-fat diet (5% of calories from carbohydrates, 30% from protein, and 65% from fat, with an energy deficit of 600 kcal/day, 3 meals distributed over 24 h: breakfast, lunch, and dinner). This intervention was performed without schedule restrictions and supported by commercial replacement meals only for the first meal (100 kcal, 15 g of protein, 3 g of fat, of which 1 g was saturated fat, and 50 mg of docosahexaenoic acid, 2 g of carbohydrates, of which < 1 g was simple sugars). After diet intervention, whole blood will be drawn and incubated with vehicle drug.
Dietary Supplement: Ketogenic diet + aspirin — The calorie-restricted KD intervention consisted of a very-low-carbohydrate, high-fat diet (5% of calories from carbohydrates, 30% from protein, and 65% from fat, with an energy deficit of 600 kcal/day, 3 meals distributed over 24 h: breakfast, lunch, and dinner). This intervention was performed without schedule restrictions and supported by commercial replacement meals only for the first meal (100 kcal, 15 g of protein, 3 g of fat, of which 1 g was saturated fat, and 50 mg of docosahexaenoic acid, 2 g of carbohydrates, of which < 1 g was simple sugars). After diet intervention, whole blood will be drawn and incubated with aspirin.

SUMMARY:
This dietary intervention study was designed to investigate the impact of a ketogenic diet on platelet function and and thrombus formation. Based on our preclinical observations, the study also aimed to discover whether aspirin could effectively counteract the ketogenic diet-induced enhancement of platelet function and attenuate the associated prothrombotic state.

DETAILED DESCRIPTION:
A randomized controlled trial was conducted to evaluate the impact of a ketogenic diet (KD) on platelet function and thrombus formation compared to a normal diet. Participants who met the specified inclusion and exclusion criteria were randomly assigned to either the KD group or the control group. The KD group followed a calorie-restricted, very-low-carbohydrate, high-fat diet for 7 days (5% carbohydrates, 30% protein, 65% fat, with a daily energy deficit of 600 kcal). To ensure compliance, one meal per day was provided as a commercial replacement. The normal diet group was instructed to maintain their original eating habits and rhythms. Whole blood was collected from the median cubital vein at baseline (pre-intervention) and after 7 days of the dietary intervention. Plasma ketone body levels were measured at both time points. To determine the effects of aspirin, the post-intervention whole blood was incubated ex vivo with either aspirin or a vehicle control. Platelet function was subsequently analyzed using platelet aggregation and ATP release assays, while thrombus formation was evaluated using a microfluidic whole-blood perfusion assay.

ELIGIBILITY:
Inclusion Criteria:

1. Participants reside in Shanghai.
2. Participants have completed Zhongshan Ketogenic Diet Study 1 in 2025.

Exclusion Criteria:

1. Pecent anti-platelet drug usage.
2. Participants with metabolic diseases including diabetes, hypertension and cardiovascular diseases.
3. Participants with craniocerebral trauma, cancer, liver disease, kidney disease, or other critical illness, or history of operation or medication.
4. Being or to be pregnant or lactating.
5. Participants with bulimia nervosa, post-traumatic stress disorder , chronic anxiety and depression or other critical neuronal disorder or history of relevant medication.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-08-18 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Platelet aggregation and ATP release | Day 8
  Platelet aggregation and ATP release were measured simultaneously using a lumi-aggregometer. Platelet aggregation was stimulated with collagen, thrombin, and ADP, while ATP release was induced by collagen and thrombin.

SECONDARY OUTCOMES:
Thrombus formation | Day 8
  Thrombus formation will be evaluated by a microfluidic whole-blood perfusion assay.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided